CLINICAL TRIAL: NCT02676219
Title: Pilot Study to Investigate the Reparative Effect of a Two Phase Oral Care Product Containing SMFP and NaF on Enamel Against a Dietary Acid Exposure Utilising an Impression Technique to Capture in Vivo Images of Teeth
Brief Title: Pilot Study Utilising an Impression Technique to Capture in Vivo Images of Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: University of Bristol Dental Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ORL-IST-2190
Record Dates: First submitted 2015-12-09; First posted 2016-02-08 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Tooth Erosion
MeSH Terms: conditions — Tooth Erosion | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RS01 (Experimental): oral care product containing containing sodium monofluorophosphate and sodium fluoride
  Interventions: Other: RS01
- Water (Placebo Comparator): Water
  Interventions: Other: Water

INTERVENTIONS:
Other: RS01 — Oral Care product containing sodium monofluorophosphate and sodium fluoride
  Arms: RS01
Other: Water
  Arms: Water

SUMMARY:
The study design is a randomised, split mouth, blind with respect to study analysts (microscopist, image grader) two treatment clinical study in 10 healthy participants with sound tooth enamel. The study will comprise of a screening visit, pre-baseline visit and 5 subsequent clinic visits. At the screening visit, participants will give consent to participate in the study. Medical history and concomitant medications will be recorded. Eligibility will be determined following an oral soft tissue (OST) examination and an evaluation of dentition exclusions. Two suitable anterior teeth will be identified for study assessments, these teeth must be at least one tooth apart in the mouth. Saliva samples will be collected from the participants at set points during the study to look at any changes in salivary pH.

ELIGIBILITY:
Inclusion Criteria:

1. Consent: Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
2. Age: Aged at least 18 years.
3. Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions.
4. General Health: Good general health with (in the opinion of the investigator or medically qualified designee) no clinically significant and relevant abnormalities of medical history or physical examination.
5. Diagnosis:

   1. Study teeth must show no signs of exposed dentine at the cervical margin.
   2. In the opinion of the investigator the study teeth must have a healthy gingiva as determined during the OST examination.

Exclusion Criteria:

1. Pregnancy Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
2. Breast-feeding Women who are breast-feeding.
3. Disease

   1. Current or recurrent disease/dental pathology that could affect the assessments.
   2. In the judgement of the investigator or medically qualified designee, any condition or medication which is causing cause Xerostomia.
   3. Diabetes Mellitus.
   4. Susceptibility to acid regurgitation.
   5. Be susceptible to high dental erosion after drinking acidic soft drinks or juices
4. General Dental Exclusions

   1. Any orthodontic appliances, restorations, bridgework or dentures that would interfere with the study evaluations or scheduled for such treatment within the timescale of the study.
   2. Recurrent or regular aphthous ulcers.
   3. Severe gingivitis, carious lesions treated and untreated periodontal disease.
   4. Excessive signs of dental erosion or a previous history of being susceptible to high dental erosion after drinking acidic drinks
   5. Tooth bleaching within past 2 months.
   6. Suffer from dentine hypersensitivity.
5. Allergy/Intolerance Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
6. Clinical Study/Experimental Medication

   1. Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
   2. Previous randomisation into this study.
7. Substance abuse Recent history (within the last year) of alcohol or other substance abuse.
8. Personnel An employee of the sponsor, member of the study site or a staff family relative. The site for this protocol is the Clinical Trials Unit in the Bristol Dental School and Hospital. Employees of the Bristol Dental School and Hospital not associated with the Clinical Trials Unit are eligible to participate.
9. Any participant who, in the judgement of the investigator, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-09-18 (Actual); Study Completion 2015-09-18 (Actual)

PRIMARY OUTCOMES:
changes in enamel surface topography using an impression methodology with scanning electron microscopy | 6 hours

SECONDARY OUTCOMES:
changes in enamel surface topography using an impression methodology with scanning electron microscopy | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicola X West, BDS, Principal Investigator — University of Bristol Dental Hospital
Locations (1):
- School of Oral and Dental Science, Bristol, United Kingdom